CLINICAL TRIAL: NCT05774223
Title: Exploring the Effects of Prefrontal iTBS on Working Memory in Healthy Participants: a Concurrent TMS/fNIRS Study
Brief Title: Prefrontal iTBS on Working Memory
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Georg Kranz, Principal Investigator, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HSEARS20200120005-03
Record Dates: First submitted 2023-03-07; First posted 2023-03-17 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Healthy
Keywords: Theta-Burst stimulation (iTBS); Functional near-infrared spectroscopy (fNIRS); Concurrent TMS/fNIRS; Working memory
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Healthy volunteers will receive iTBS two times with active or sham stimulation separated by one week to investigate the effect duration of iTBS on working memory
Who Masked: Participant
Masking Description: Participants will not be informed of the type of stimulation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active iTBS on working memory (Active Comparator): Participants will receive active 80% rMT iTBS over the left DLPFC in this arm. The working memory assessments will be performed pre-stimulation and at 0-, 10-, 20-, 30-, and 40-min post-stimulation. The working memory assessment is measured using a 2-minute 3-back task. The fNIRS will monitor the prefrontal hemoglobin change throughout the whole procedure.
  Interventions: Device: Transcranial magnetic stimulation (TMS)-active
- Sham iTBS on working memory (Sham Comparator): Participants will receive sham 80% rMT iTBS over the left DLPFC (by putting the coil perpendicular to the left DLPFC) in this arm. The working memory assessments will be performed pre-stimulation and at 0-, 10-, 20-, 30-, and 40-min post-stimulation. The working memory assessment is measured using a 2-minute 3-back task. The fNIRS will monitor the prefrontal hemoglobin change throughout the whole procedure.
  Interventions: Device: Transcranial magnetic stimulation (TMS)-sham

INTERVENTIONS:
Device: Transcranial magnetic stimulation (TMS)-active — Active intermittent TBS (iTBS) will be applied to the left DLPFC at 80% of the resting motor threshold (rMT) (Hoy et al., 2016). A stimulation, where 3-pulse at 50 Hz will be given, will repeat every 10 s for a total of 190 s (600 pulses in total) (Huang et al., 2005). The left DLPFC stimulation site will be determined using the neuronavigator system (lDLPFC, x-38, y+44, z+26).
  Arms: Active iTBS on working memory
Device: Transcranial magnetic stimulation (TMS)-sham — Sham intermittent TBS (iTBS) will be applied to the left DLPFC at 80% of the resting motor threshold (rMT) (Hoy et al., 2016). The coil will be placed perpendicular to the left DLPFC. A stimulation, where 3-pulse at 50 Hz will be given, will repeat every 10 s for a total of 190 s (600 pulses in total) (Huang et al., 2005). The left DLPFC stimulation site will be determined using the neuronavigator system (lDLPFC, x-38, y+44, z+26).
  Arms: Sham iTBS on working memory

SUMMARY:
The investigators previous pilot study showed that the brain remained activated after 3 minutes of intermittent theta burst stimulation (iTBS). Therefore, an open question remains that how long the effects will last and when the maximum effects will be achieved. In addition, many pioneering works showed the positive effects of repetitive transcranial magnetic stimulation (rTMS) on working memory. Intermittent theta burst stimulation (iTBS) is a patterned form of rTMS, it has shown a non-inferior efficacy in depression but with a much shorter time (approximately 3 mins) than traditional rTMS (approximately 40 mins).

As discussed above, this study aims to investigate the effects of prefrontal iTBS on working memory using concurrent iTBS/fNIRS and to explore the duration of the effects.

ELIGIBILITY:
Inclusion Criteria:

* right-handed participants
* normal or corrected-to-normal vision

Exclusion Criteria:

* a current or past diagnosis of any neurological or psychiatric disorder
* any severe medical conditions, seizure, and pregnancy
* contraindication to TMS (e.g., with mental implants)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
N-back | before and post iTBS, up to 3 months
  The accuracy number of each n-back task
N-back | before and post iTBS, up to 3 months
  The response time of each n-back task

SECONDARY OUTCOMES:
Hemoglobin change | before and post iTBS, up to 3 months
  The hemoglobin change throughout whole procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No